CLINICAL TRIAL: NCT01523860
Title: Brief Induction Chemoimmunotherapy With Rituximab + Bendamustine + Mitoxantrone Followed by Rituximab in Elderly Patients With Advanced Stage Previously Untreated Follicular Lymphoma
Brief Title: Brief Chemoimmunotherapy With R+B+M Followed by R in Elderly Patients Advanced Stage Untreated Follicular Lymphoma
Acronym: FLE09
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Collaborators: Centro di Riferimento per l'Epidemiologia e la Prev. Oncologica Piemonte (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIL_FLE09
Record Dates: First submitted 2011-06-23; First posted 2012-02-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab; Mitoxantrone; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Rituximab will be supplied as 375 mg/sqm for i.v.administration.Mitoxantrone will be supplied as 8 mg/sqm for i.v.administration.Bendamustine will be supplied as 90 mg/sqm for i.v.administration.
  Interventions: Drug: Rituximab, Mitoxantrone, Bendamustine

INTERVENTIONS:
Drug: Rituximab, Mitoxantrone, Bendamustine — Rituximab will be supplied as 375 mg/sqm for i.v.administration.Mitoxantrone will be supplied as 8 mg/sqm for i.v.administration.Bendamustine will be supplied as 90 mg/sqm for i.v.administration

SUMMARY:
This is a prospective, multicenter phase II trial designed to determine efficacy and safety of a brief chemoimmunotherapy with the combination of Rituximab + Bendamustine + Mitoxantrone in elderly patients with advanced stage Follicular Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven diagnosis of B-cell CD20+ follicular NHL, grade I, II and IIIa of WHO Classification
* Untreated patients with the exception of prior limited radiotherapy
* Stage III or IV who require therapy according to SIE and GELF criteria
* Stage II with at least one of the following:

  * Bulky disease (>7 cm)
  * LDH >normal
  * Systemic symptoms
  * Beta2-Microglobulin >3 mg/l
  * Extra-nodal involvement
  * Active disease with rapid progression 5.Age from 65 to 80 years, geriatric score "FIT" (see Appendix B) 6.Life expectancy >6 months 7.ECOG performance status 0-2 (see Appendix C) 8.LVEF ≥45% or FS ≥37% 9.ANC ≥1 x 109/l and Platelets count ≥75 x 109/l, unless due to bone marrow involvement by follicular lymphoma 10.Creatinine up to 1.5 x ULN 11.Conjugated bilirubin up to 2 x ULN 12.Alkaline phosphatase and transaminases up to 2 x ULN 13.Sending of bone marrow sample for Bcl-2/IgH rearrangement evaluation 14.Written informed content

Exclusion Criteria:

* Men not agreeing to take adequate contraceptive precautions during and for at least 6 months after cessation of therapy
* History of other malignancies within 3 years prior to study entry except for: adequately treated carcinoma in situ of the cervix; basal or squamous cell skin cancer; low grade, early stage, localized prostate cancer treated surgically with curative intent; good prognosis DCIS of the breast treated with lumpectomy alone with curative intent
* Medical condition requiring long term use (>1 months) of systemic corticosteroids
* Active bacterial, viral, or fungal infection requiring systemic therapy 5. Concurrent medical condition which might exclude administration of therapy
* Cardiac insufficiency (NYHA grade III/IV; see Appendix D)
* Myocardial infarction within 6 months of entry on study
* Severe chronic obstructive pulmonary disease with hypoxemia
* Severe diabetes mellitus difficult to control with adequate insulin therapy
* Hypertension that is difficult to control
* Impaired renal function with creatinine clearance <30 ml/min (see Appendix E)
* HIV positivity
* HBV positivity with the exception of patients HbsAg negative and Ab anti-Hbcore positive (these patients need to receive prophylaxis with Lamivudine)
* HCV positivity with the exception of patients with no laboratory signs of active chronic hepatitis and HCV-RNA negativity
* CNS involvement by lymphoma 16. Participation at the same time in another study in which investigational drugs are used
* Known hypersensitivity or anaphylactic reactions to murine antibodies or proteins
* Any other co-existing medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Complete Response (CR) Rate at the end of the consolidation phase | 6 months
  Proportion of CR according to the Cheson 2007 response criteria

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 24 months
  PFS will be measured from the day of enrolment to the date of disease progression, relapse or death due to any cause.
Molecular response rate (Bcl2/IgH rearrangement) | 24 months
  Rate of conversion to molecular remission by qualitative and quantitative PCR only in patients with a positive marker at baseline
Molecular relapse rate | 24 moths
  Rate of conversion to molecular relapse measured by PCR only in patients with a positive marker at baseline
Incidence of grade 3 or greater overall toxicities measured by CTCAE v.3.0 | 24 months
Overall survival (OS) | 24 moths
  OS will be measured from the day of enrolment to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Vitolo, MD, Study Director — Azienda Sanitaria Ospedaliera-Universitaria S. Giovanni Battista - TORINO
Locations (37):
- Italy (37):
  - Divisione di Ematologia Ospedale SS. Antonio e Biagio, Alessandria, Alessandria
  - SOS Ematologia Ospedale C. Massaia, Asti, Asti
  - Ematologia con Trapianto, Università di Bari, Bari, Bari
  - Medicina Interna, Ospedale degli Infermi, Biella, Biella
  - Istituto di Ematologia ed Oncologia Medica A. Seragnoli Policlinico S. Orsola, Bologna, Bologna
  - Divisione di Ematologia e TMO, Ospedale di Bolzano, Bolzano, Bolzano
  - S.C. di Ematologia, Spedali Civili, Brescia, Brescia
  - Divisione di Ematologia, Ospedale Businco, Cagliari, Cagliari
  - Divisione di Ematologia, Ospedale di Catania, Catania, Catania
  - Azienda Ospedaliera Santa Croce e Carle, Cuneo, Cuneo
  - Clinica Ematologica Policlinico Carreggi, Florence, Firenze
  - Divisione di Ematologia, Policlinico Careggi, Florence, Firenze
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.), Meldola, Forlì-Cesena
  - Ematologia I, A.O.U. San Martino, Genova, Genova
  - Ematologia e Trapianto Ospedale Card.Panico, Tricase, Lecce
  - S.C. Ematologia, Azienda Ospedaliera Papardo, Messina, Messina
  - Divisione di Ematologia, Ospedale Niguarda, Milan, Milano
  - Ematologia e Trapianto IRCCS, Istituto Nazionale dei Tumori, Milan, Milano
  - Policlinico La Marcora, Milan, Milano
  - Ematologia, A.O. San Gerardo, Monza, Milano
  - Oncologia Medica ed Ematologia, Istituto Clinica Humanitas, Rozzano, Milano
  - UO Ematologia, II Facoltà di Medicina e Chirurgia Università Federico II, Napoli, Napoli
  - SCDU Ematologia, AOU Maggiore della Carità, Novara, Novara
  - UO Ematologia, Università - Policlinico San Matteo, Pavia, Pavia
  - Divisione di Oncologia Medica A, Centro di Riferimento Oncologico, Aviano, Pordenone
  - Ematologia Ospedale Santa Maria delle Croci, Ravenna, Ravenna
  - Div. Ematologia A.O. "Bianchi Melacrino Morelli", Reggio Calabria, Reggio Calabria
  - UO Oncologia ed Onco-Ematologia, Ospedale di Rimini, Rimini, Rn
  - Università Cattolica del Sacro Cuore, Roma, Roma
  - Dipartimento di biotecnologie cellulari ed ematologia Ospedale Umberto I, Università La Sapienza, Roma, Roma
  - Ospedale Santa Maria di Terni, Terni, Terni
  - Osp. San Giovanni Battista - Biologia Molecolare, Torino, Torino
  - Osp. San Giovanni Battista - Ematologia 2, Torino, Torino
  - Ospedale S. Chiara, Trento, Trento
  - Ematologia Ospedale Santa Maria Di Ca' Foncello, Treviso, Treviso
  - Clinica di Ematologia, A.O.U. di Udine, Udine, Udine
  - S.C. Medicina Trasfusionale ed Ematologia , P.O. Ivrea, Ivrea

REFERENCES:
- [Derived] Boccomini C, Ladetto M, Rigacci L, Puccini B, Rattotti S, Volpetti S, Ferrero S, Chiarenza A, Freilone R, Novo M, Corradini P, Nassi L, Rusconi C, Stelitano C, Bolis S, Marina Liberati A, Tucci A, Baldini L, Balzarotti M, Evangelista A, Ciccone G, Vitolo U. A brief rituximab, bendamustine, mitoxantrone (R-BM) induction followed by rituximab consolidation in elderly patients with advanced follicular lymphoma: a phase II study by the Fondazione Italiana Linfomi (FIL). Br J Haematol. 2021 Apr;193(2):280-289. doi: 10.1111/bjh.17283. Epub 2021 Jan 21. PMID 33476434